CLINICAL TRIAL: NCT03097952
Title: "Real-life" Cohort Study on Patients With Chronic Hepatitis B Virus Infection in Jiangsu
Brief Title: "Real-life" Cohort Study on Patients With Chronic HBV Infection in Jiangsu
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Chao Wu, Prof., The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: NJDTID-001
Record Dates: First submitted 2017-03-06; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B， Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy tissue, blood (serum, plasma, and DNA)

SUMMARY:
Hepatitis B virus (HBV) infection remains one of the most serious health problems worldwide. Patients with chronic HBV infection are at an increased risk for developing hepatic cirrhosis, hepatocellular carcinoma and even death. Although some predictive factors of the outcome of chronic HBV infection were identified, more precisely determine the factors which are associated with the outcome in non-selected patients with chronic HBV infection are still needed. The investigators purpose is to constitute a observational cohort of non-selected Chinese patients to create a database of epidemiological, clinical, biological, virological, immunologic and therapeutic parameters, in order to determine factors associated with the outcome of chronic HBV infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic HBV infection (defined as HBsAg positive for at least 6 months)

Exclusion Criteria:

* Co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) and/or hepatitis D virus (HDV)
* History of liver transplantation
* History of hepatocellular carcinoma (HCC)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients chronically infected with hepatitis B virus
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2008-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with antigen loss (HBeAg and HBsAg loss) | 20 years
Cirrhosis | 20 years
Hepatic decompensation | 20 years
  Development of hepatic decompensation will be defined by any of the following events:
  (1) Ascites or hepatic hydrothorax; (2)Variceal or portal hypertensive bleeding; (3)Hepatic encephalopathy
Hepatocellular carcinoma (HCC) | 20 years
  The diagnosis of HCC will be made using the American Association for the Study of Liver Disease criteria.
Death | 20 years
  Date and cause of death will be recorded.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The Third Hospital of Changzhou, Changzhou, Jiangsu
  - Huai'an No.4 People's Hospital, Huai'an, Jiangsu
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nanjing Jiangbei People's Hospital, Nanjing, Jiangsu
  - Suqian People's Hospital, Suqian, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu

REFERENCES:
- [Derived] Wang J, Zhu L, Zhang Z, Zhang S, Pan Y, Li Y, Cao F, Jiang C, Fan T, Xiong Y, Liu J, Chen Y, Yin S, Tong X, Zhu C, Liu X, Li J, Wu C, Huang R. Lower HBV DNA level is associated with more severe liver fibrosis in HBeAg-positive chronic hepatitis B with normal alanine transaminase. Virol J. 2024 Jun 4;21(1):127. doi: 10.1186/s12985-024-02368-0. PMID 38835029
- [Derived] Yao R, Lu S, Xue R, Wang J, Qiu Y, Chen Y, Liu J, Zhu L, Zhan J, Jiang S, Yin S, Tong X, Ding W, Li J, Zhu C, Huang R, Wu C. NAFLD is associated with less severe liver fibrosis in chronic hepatitis B: A multi-center, retrospective study. Ann Hepatol. 2024 Jan-Feb;29(1):101155. doi: 10.1016/j.aohep.2023.101155. Epub 2023 Sep 24. PMID 37742745
- [Derived] Wang J, Liu J, Liu Y, Xue R, Zhan J, Jiang S, Wang L, Yan X, Xiong Y, Xia J, Yin S, Tong X, Chen Y, Li J, Huang R, Wu C. Clinical features of chronic hepatitis B patients with lean nonalcoholic fatty liver disease. Hepatol Res. 2023 Mar;53(3):184-195. doi: 10.1111/hepr.13854. Epub 2022 Nov 21. PMID 36317959